CLINICAL TRIAL: NCT02061735
Title: Ontogeny and Quantitative Multimodal Skin Imaging of Infantile Hemangiomas
Brief Title: Ontogeny of Infantile Hemangiomas With Skin Imaging Modalities
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Society for Pediatric Dermatology (Other)
Responsible Party: Sponsor
Other Study IDs: CHMC 2011-0443
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Infantile Hemangiomas
Keywords: skin imaging; image analysis; infrared thermography; infantile hemangioma; three dimensional imaging; color imaging and analysis; propranolol; timolol; ontogeny
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- oral propranolol: Dosage of 1 mg/kg per day divided 2 times daily. Blood pressure, heart rate and oxygen saturation are monitored after propranolol initiation. Treatment is continued with a gradual increase to 2 mg/kg per day divided 2 times daily. Treatment is continued until the hemangioma no longer changes in the characteristics judged by the physicians, including, color, size, temperature and deformability.
- timolol maleate 0.5% gel: One drop of of timolol maleate 0.5% gel is topically applied and massaged into the hemangioma twice per day . This dosage provides an estimated 0.5 mg of timolol per day. The treatment is continued until it is considered to be no longer effective as judged by the physicians.
- No treatment, observation only: No oral or topical treatment will be given as recommended by the treating physicians and elected by the parents. Patients will be evaluated periodically to determine what changes in treatment are warranted. If this occurs, the patients will be included in the appropriate study group.

SUMMARY:
A combined set of quantitative skin imaging methods will quantitatively describe the natural ontogeny and the response to standard treatments over time in patients with infantile hemangiomas.

DETAILED DESCRIPTION:
Infantile hemangiomas (IH) are relatively common benign vascular neoplasms, which appear shortly after birth and grow rapidly in the following weeks and months. The proliferative phase involves a rapidly dividing endothelial cell proliferation. The tumors generally stabilize and then involute over time. They are usually clinically insignificant; however, a small percentage of them can be life threatening secondary to location, associated syndrome, and physical findings such as ulceration. Treatment options have included steroids, interferon, vincristine and more recently propranolol. There are few published prospective research studies on the effectiveness of these treatment options. Because of several factors, it has been difficult to objectively measure response of these lesions. The purpose is to determine (1) whether multiple quantitative skin imaging modalities can quantitatively describe the clinically relevant features of infantile hemangiomas, including color (red, blue), lightness, size (height, volume), biomechanical properties, temperature and perfusion and (2) the natural ontogeny and response to treatment over time. The treatments are oral propranolol, topical timolol and untreated (observation).

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 5 years of age
* Diagnosis of a cutaneous infantile hemangioma
* Diagnosis of hemangioma requiring treatment (treatment includes: propranolol or topical timolol) or diagnosis of an infantile hemangioma that will not be treated at the time of enrollment
* Able to tolerate imaging procedures

Exclusion Criteria:

* Age > 5 years
* Non cutaneous infantile hemangioma
* Hemangioma on the lip
* Hemangioma on the eyelid
* Hemangioma located in areas whereby measurements cannot be made due to equipment limitations
* Deep hemangioma with no visible skin surface component
* Congenital hemangioma
* No available normal site for study control
* Other vascular anomaly
* Not able to tolerate imaging procedures

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients being seen at the the Hemangioma and Vascular Malformation Center of Cincinnati Children's Hospital Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hemangioma height | up to 5 years
  IH height and volume will be obtained from surface scans with the Artec scanner with a 0.5 mm resolution, 0.1 mm accuracy, at 60 cm. Three dimensional scans will be created with the Artec Studio software and features quantified with the three dimensional software. Soft tissue landmarks will create the region of interest for all evaluations. Height and volume will be calculated for the infantile hemangioma versus the control.
Static and Dynamic Temperature | up to 5 years
  Temperature information will be acquired with a thermal imaging camera with analysis software. The thermal features of the surrounding uninvolved control skin are removed by applying thresholds. Static infrared thermography captures the steady-state condition and spatial distribution. Dynamic infrared thermography applies a stress (cooling) to stimulate the thermal response within the tissue.
Skin color and lightness | up to 5 years
  High resolution color Images will be taken taken with a digital camera, Micro 60 mm lens with a wireless close up flash system at 30cm and perpendicular to the site. The images are color corrected and processed into three distinct images : red color, blue-yellow color, and lightness (white - back).
  Color and thermal images are co-registered and analyzed with customized software. The system creates quantitative outputs and maps for visualization of IH regions of thermal and color activity. Threshold values for the lightness, red color, blue color and thermal images are selected based upon histogram distributions of the uninvolved skin as the values above the mean and multiple standard deviations The pixels beyond the thresholds are used to quantify and map the features due to the hemangioma itself.

SECONDARY OUTCOMES:
Biomechanical properties | up to 5 years
  Tissue mechanical properties (i.e., elasticity, elastic deformation, laxity, stiffness, etc.) will be measured to assess tissue deformability. The instrument measures biomechanical properties of the skin by applying a negative pressure, in the range between 20 and 500 mbar. These properies are compared to an uninvolved contralateral control site.

CONTACTS AND LOCATIONS:
Overall Officials: Marty O Visscher, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Denise Adams, MD, Study Chair — Children's Hospital Medical Center, Cincinnati; Adrienne Hammill, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Burkes SA, Patel M, Adams DM, Hammill AM, Eaton KP, Randall Wickett R, Visscher MO. Infantile hemangioma status by dynamic infrared thermography: A preliminary study. Int J Dermatol. 2016 Oct;55(10):e522-32. doi: 10.1111/ijd.13298. Epub 2016 Apr 8. PMID 27062495